CLINICAL TRIAL: NCT03167099
Title: Immediate Weight Bearing as Tolerated Versus Protected Weight Bearing in Supracondylar Distal Femur Fractures; a Prospective, Randomized Study
Brief Title: Immediate Weight Bearing Versus Protected Weight Bearing in Supracondylar Distal Femur Fractures
Acronym: WtBrFemFx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, David Hubbard, MD, MD, Chief, Orthopaedic Trauma Service, Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1408401969A
Record Dates: First submitted 2015-04-08; First posted 2017-05-25 (Actual); Results first posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-06

CONDITIONS: Closed Supracondylar Fracture of Femur

STUDY DESIGN:
Masking Description: Both investigators and participants are aware of the assignment. There is no masking; only randomization.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Full Weight Bearing (Experimental): Participants assigned to full weight bearing after fixation of distal femur fracture.
  Interventions: Procedure: Full Weight Bearing
- Partial Weight Bearing (No Intervention): Participants assigned to partial weight bearing, standard of care, after fixation of distal femur fracture.

INTERVENTIONS:
Procedure: Full Weight Bearing — full weight bearing after fixation of a distal femur fracture
  Arms: Full Weight Bearing

SUMMARY:
This study is designed to examine if immediate weight bearing on a distal femur fracture fixed with a primary locking plate, either a distal condylar locking plate or a LISS (less invasive stabilization system), is safe and promotes more rapid fracture healing than partial weight bearing, which is standard of care.

DETAILED DESCRIPTION:
This study is designed to examine if immediate weight bearing on a distal femur fracture fixed with a primary locking plate, either a distal condylar locking plate or a LISS (less invasive stabilization system), is safe and promotes more rapid fracture healing than partial weight bearing, which is standard of care. Historically and currently patients are kept partial weight bearing after fixation of these fractures for 6-12 weeks until callous formation is observed on radiographs. The hypothesis is that participants allowed to bear weight immediately will heal at least as quickly as those who have weight bearing status protected with the added benefits from early mobilization. Fracture healing will be monitored closely by follow up appointments and complications will be documented.

ELIGIBILITY:
Inclusion Criteria:

* aged > 18 yo
* distal supracondylar femur fracture (Supracondylar distal femur fractures treated with a locked plate, either a distal condylar locking plate or a LISS (less invasive stabilization system), including peri-prosthetic fractures)
* both male and female

Exclusion Criteria:

* Patients with an intracondylar split,
* polytrauma patients with associated trauma that will inhibit their ability to weight bear,
* metastatic disease,
* incomplete follow up,
* subjects with questionable ability to bear weight (ie advanced dementia),
* open fractures with bone loss.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David F Hubbard, MD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers. Shared group data will be presented at Orthopaedic conferences and through manuscript submission.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Full Weight Bearing | Partial Weight Bearing
Started | 26 | 27
Completed | 19 | 19
Not Completed | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Full Weight Bearing: Participants assigned to full weight bearing after fixation of distal femur fracture.
  Full Weight Bearing: Participants will be randomized to one of two groups; full weight bearing, which is the intervention, or partial weight bearing, which is standard of care, after fixation of a distal femur fracture.
- Total: Total of all reporting groups
Arm/Group | Full Weight Bearing | Partial Weight Bearing | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 10
  >=65 years | 22 | 21 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 47
  Male | 3 | 3 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Time to Distal Femur Fracture Healing by Radiographic Evidence
Description: Radiographs were analyzed postoperatively to determine bridging of 3 or 4 cortices per standard of care during follow-up office visits.
Time Frame: up to 12 weeks
Population: Radiographic evidence not available for 4 subjects in each arm.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Full Weight Bearing | Partial Weight Bearing
Number analyzed (Participants) | 22 | 23
months | 1.75 (0.63) | 2.15 (0.87)

2. Secondary Outcome: Time to Ambulation
Description: Investigators measure time to ambulation
Time Frame: up to 24 weeks
Population: Time to ambulation not collected for 7 participants in full weight bearing group; 8 participants in partial weight bearing group
Measure: Mean (Full Range); unit: Weeks
Arm/Group | Full Weight Bearing | Partial Weight Bearing
Number analyzed (Participants) | 19 | 19
Weeks | 9.947 [0 to 24] | 15.316 [6 to 24]

3. Secondary Outcome: Time of Participation in Physical Therapy
Description: Investigators measure the length of time of physical therapy participation
Time Frame: up to 1 year
Population: Data was not collected.
Arm/Group | Full Weight Bearing | Partial Weight Bearing
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Number of Days to Discharge
Description: Investigators record the number of days from surgery to discharge
Time Frame: Up to 30 days
Measure: Mean (Full Range); unit: Days
Arm/Group | Full Weight Bearing | Partial Weight Bearing
Number analyzed (Participants) | 26 | 27
Days | 6.115 [2 to 23] | 6.074 [2 to 17]

5. Other Pre Specified Outcome: Discharge Disposition
Description: Investigators record the participants' discharge location, e.g. home, rehabilitation facility
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Full Weight Bearing | Partial Weight Bearing
Number analyzed (Participants) | 26 | 27
Participants
  Home | 5 | 5
  Skilled Nursing Facility | 10 | 18
  Acute Rehab | 10 | 4
  Hospice/Comfort Measures Only | 1 | 0

6. Other Pre Specified Outcome: Change in Pain
Description: Investigators record the pain from 0-10 at each time point
Time Frame: 2 days, 2 weeks, 6 weeks, 3 months, 6 months, 12 months
Population: Data was not collected.
Arm/Group | Full Weight Bearing | Partial Weight Bearing
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Change in Knee Society Score
Description: Participants complete the Knee Society survey at the listed time points
Time Frame: 6 weeks, 3 months, 6 months, 12 months
Population: Data not collected.
Arm/Group | Full Weight Bearing | Partial Weight Bearing
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Knee Flexion
Description: Investigators measure knee flexion
Time Frame: 12 months
Population: Knee flexion was not measured in 3 subjects in the full weight bearing group and 5 subjects in the partial weight bearing group.
Measure: Mean (Full Range); unit: Degrees
Arm/Group | Full Weight Bearing | Partial Weight Bearing
Number analyzed (Participants) | 23 | 22
Degrees | 101 [40 to 130] | 97 [70 to 130]

9. Other Pre Specified Outcome: Number of Participants With Non Union
Description: Investigators assess non union at 1 year
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Full Weight Bearing | Partial Weight Bearing
Number analyzed (Participants) | 26 | 27
Participants | 0 | 3

10. Other Pre Specified Outcome: Number of Participants With Malunion
Description: Investigators assess malunion at 1 year
Time Frame: 12 months
Population: Data was not collected.
Arm/Group | Full Weight Bearing | Partial Weight Bearing
Number analyzed (Participants) | 0 | 0

11. Other Pre Specified Outcome: Number of Participants With Infection
Description: Investigators check for infection
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Full Weight Bearing | Partial Weight Bearing
Number analyzed (Participants) | 26 | 27
Participants | 0 | 1

12. Other Pre Specified Outcome: Deep Vein Thrombosis at Each Time Point
Description: Investigators check for Deep Vein Thrombosis
Time Frame: 12 months
Population: Data was not collected.
Arm/Group | Full Weight Bearing | Partial Weight Bearing
Number analyzed (Participants) | 0 | 0

13. Other Pre Specified Outcome: Number of Participants With Pulmonary Embolism
Description: Investigators check for Pulmonary Embolism
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Full Weight Bearing | Partial Weight Bearing
Number analyzed (Participants) | 26 | 27
Participants | 0 | 1

14. Other Pre Specified Outcome: Number of Participants With Implant Failure
Description: Investigators check for implant failure at 12 months
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Full Weight Bearing | Partial Weight Bearing
Number analyzed (Participants) | 26 | 27
Participants | 2 | 2

15. Other Pre Specified Outcome: Change in Vit D Level in Age 65 and Older
Description: Investigators assess Vit D level in subject age 65 and older at all time points listed
Time Frame: baseline, 2 weeks, 6 weeks, 3 months, 6 months, 12 months
Population: Data was not collected.
Arm/Group | Full Weight Bearing | Partial Weight Bearing
Number analyzed (Participants) | 0 | 0

16. Other Pre Specified Outcome: Study Mortality
Description: Investigators record any deaths at 12 months
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Full Weight Bearing | Partial Weight Bearing
Number analyzed (Participants) | 26 | 27
Participants | 3 | 7

ADVERSE EVENTS:
Time Frame: 1 year from date of surgery
Description: Charts were reviewed at every clinic visit post operatively.
Arm/Group | Full Weight Bearing | Partial Weight Bearing
All-Cause Mortality (participants affected / at risk) | 3/26 | 7/27
Serious Adverse Events (participants affected / at risk) | 2/26 | 2/27
Other Adverse Events (participants affected / at risk) | 0/26 | 1/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full Weight Bearing (N=26) | Partial Weight Bearing (N=27)
Failure of Fixation (Product Issues) | 1 (1) | 0 (0) — X-ray shows failure of fixation of right distal femur fracture. Removal of hardware with right distal femoral replacement performance
Fracture from fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Fell day after discharge following initial femur repair, fracturing other side. ORIF (open reduction and internal fixation) to other femur performed.
Nonunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Evidence of left distal femoral nonunion. Revision performed 11 months postoperatively.
Fall unknown source (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Left periprosthetic proximal femur fracture, open exam under anesthesia performed.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full Weight Bearing (N=26) | Partial Weight Bearing (N=27)
COPD (Chronic Obstructive Pulmonary Disease) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Visit to Emergency Department, complaints of shortness of breath and back pain. Chest x-ray, EKG, and lab work were completed. Clinically stable and discharged home same day. Instructed to follow-up with primary care provider.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT03167099/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT03167099/ICF_001.pdf